CLINICAL TRIAL: NCT07218159
Title: Can an Evidence-based Sexual Assault Resistance Intervention Also Prevent Intimate Partner Violence (IPV)? A Randomized Controlled Trial Sub-Study of the Efficacy of IDEA3 for Reducing IPV in Undergraduate Women
Brief Title: Can the IDEA3 Intervention Prevent Intimate Partner Violence?: A Substudy to the IDEA3 Randomized Controlled Trial
Acronym: IDEA3-IPV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Windsor (Other); University of Guelph (Other); University of Central Florida (Other); University of Michigan (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Sarah Peitzmeier, Associate Professor of Behavioral and Community Health, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB# 23-063
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Intimate Partner Violence (IPV)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDEA3 sexual assault resistance intervention (Experimental): IDEA3 curriculum will be delivered by pairs of trained facilitators over Zoom to reach up to 8 pairs of female-identified university students in four, 3-hour units. The four units will be spread over two to four weeks' time.
  Interventions: Behavioral: IDEA3 Sexual Assault Resistance Intervention
- Consent workshop (Active Comparator): Randomized participants who do not receive the intervention will receive one 60-minute session consisting of an internet delivered (Zoom) consent workshop.
  Interventions: Behavioral: Consent workshop

INTERVENTIONS:
Behavioral: IDEA3 Sexual Assault Resistance Intervention — Internet-delivered EAAA (IDEA3), adapted from an in-person sexual assault resistance education intervention: Enhanced Assess, Acknowledge, Act (EAAA) intervention that was found in a randomized trial to reduce sexual assault victimization by about 50% at follow-up. IDEA3 designed for female identifying university students and focuses on resisting sexual assault committed by males in 4, 3-hour units: 1-ASSESS builds ability to detect risk with male acquaintances and develop risk reduction strategies. 2-ACKNOWLEDGE explores overcoming emotional barriers preventing women from acknowledging risk and employing effective resistance strategies with males. 3-ACT shows effectiveness of resistance strategies and teaches verbal and physical self-defense in common situations. 4-RELATIONSHIPS & SEXUALITY adapts the Our Whole Lives curriculum to increase women's comfort in talking about sex/sexuality and identify sexual values/desires.
  Arms: IDEA3 sexual assault resistance intervention
Behavioral: Consent workshop — Participant pairs assigned to the control arm will receive a 60-minute session consisting of a 60-min interactive, virtual consent workshop. The workshop will include information on a) what consent is, including the idea that consent is about bodily autonomy and applies to interactions beyond sex, b) how to give and ask for consent, and c) examples of what it looks like to ask for and give/not give consent. This presentation will be given by a well-trained Research Assistant.
  Arms: Consent workshop

SUMMARY:
The goal of this study is to understand if the Internet-Delivered Enhanced Assess, Acknowledge, Act (IDEA3) sexual assault resistance program works to prevent intimate partner violence in undergraduate women. Participants who were in a prior trial by the study team (the IDEA3 parent trial) and joined in September 2024 or later will be invited to also join this study at the conclusion of the parent study. Participants in this study will fill out one additional survey. Researchers will compare intimate partner violence victimization between the control group and the intervention group.

DETAILED DESCRIPTION:
About 1 in 4 undergraduate women experience intimate partner violence (IPV) before graduation, and 1 in 5 women experience sexual assault (SA). IPV and SA are linked to academic or professional consequences for women who are victimized in college, including decreased class attendance, difficulty concentrating on schoolwork, withdrawing from classes, and dropping out of higher education entirely. The Enhanced Assess, Acknowledge, Act (EAAA) program is the only intervention proven to reduce the one-year incidence of campus SA in a randomized controlled trial (RCT) by 50%. A trial sub-study showed that EAAA also reduced IPV victimization by over 50%. EAAA is a theory-based 12-hour group intervention that increases women's abilities to assess a situation (cognitive appraisal to recognize empirically supported "red flags"), quickly acknowledge the potential for assault (e.g., overcoming self-doubt that one may be misreading the situation), and act to resist SA using evidence-based strategies. However, uptake of this effective in-person program has been limited by the cost and burden for college campuses to implement the program themselves. The researchers are currently testing an online adaptation of EAAA known as Internet-Delivered EAAA (IDEA3) in a Canadian-funded RCT, to evaluate a version of EAAA that will be more feasible to implement widely. An online format would lower costs and allow a central non-profit to deliver the program nationwide, with students from any campus participating via Zoom. While the trial was designed to evaluate the effect of IDEA3 on SA, the researchers will add an IPV sub-study to the trial. This sub-study will determine the efficacy of IDEA3 in reducing the one-year incidence of IPV, as compared to a consent workshop control condition, in US undergraduate women. The results of the study will provide key data that can be used to scale an evidence-based solution to this critical and timely issue.

This is an add-on sub-study to NCT06058455. Participants recruited in September 2024 and later into NCT06058455 will be invited to participate in this sub-study at their 12-month survey. Participants will be invited to fill out a survey on experiences of intimate partner violence (IPV) over the prior 12 months. This sub-study will enable us to determine the efficacy of IDEA3 in reducing the one-year incidence of IPV, as compared to a consent workshop control condition, in undergraduate women.

ELIGIBILITY:
Inclusion Criteria: Enrolled in the IDEA3 parent study in September 2024 or later and completed the 12 month survey for the parent trial

Original inclusion criteria for the parent trial:

* 1st- and 2nd-year university students at one of the 4 sites
* female-identifying students
* students between ages of 17-24 at the time of enrollment into the parent trial
* able to attend one of the scheduled program groups
* able and willing to be matched with another eligible student

Exclusion Criteria:

* None

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender or transgender women
Enrollment: 289 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Physical and psychological intimate partner violence | 12 months
  The Composite Abuse Scale Revised-Short Form (CASR-SF) will be used to measure IPV. The scale will be administered as written (16 items), but two questions relating to sexual IPV are removed from the scale in analysis to avoid overlap with sexual assault as an outcome. Thus, the modified CASR-SF uses 14 questions to measure physical and psychological IPV. Participants indicate the frequency with which they experienced each item, from never (0) to daily (5) and are determined to have experienced IPV based on validated cutoffs. All occurrences of IPV in all new relationships since the participants' enrollment in the main IDEA3 trial will be recorded. If a participant had multiple relationships, they will be asked to indicate in which relationship(s) the IPV had occurred.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - University of Central Florida, Orlando, Florida
  - University of Maryland, College Park, Maryland
  - University of Michigan, Ann Arbor, Michigan
- Canada (2):
  - University of Guelph, Guelph, Ontario
  - University of Windsor, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Qualified academic researchers will be allowed to access de-identified survey responses upon request to the PIs, or a designee such as a secure data repository, e.g. ICPSR. The final system for managing and approving requests has yet to be determined.
Supporting Information: Study Protocol, SAP
Time Frame: From first publication and available for at least 5 years
Access Criteria: The final system for managing and approving requests has yet to be determined.